CLINICAL TRIAL: NCT01719770
Title: Requirement of Skeletal Muscle Paralysis in Hypothermic Patients After Cardiac Arrest - a Pilot Study
Brief Title: Skeletal Muscle Paralysis in Hypothermic Patients After Cardiac Arrest
Acronym: RELAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Heidrun Losert, Priv. Doz. Dr. Heidrun Losert, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RELAX1
Record Dates: First submitted 2011-07-06; First posted 2012-11-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Cardiac Arrest With Successful Resuscitation; Hypothermia; Skeletal Muscle Relaxant Overdose
Keywords: cardiac arrest; therapeutic hypothermia; skeletal muscle paralysis; shivering; serum drug levels; basal metabolism
MeSH Terms: conditions — Hypothermia; Heart Arrest | interventions — Rocuronium; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rocuronium (Active Comparator): Continuous infusion of rocuronium with 0,25mg/kg (blinded) for 29 hours after initiation of mild therapeutic hypothermia
  Interventions: Drug: rocuronium
- Placebo (Placebo Comparator): Continuous infusion of sodium-chloride (placebo) and rocuronium bolus (0,25mg/kg)in case of shivering episode (blinded)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: rocuronium — continuous application of rocuronium 0,25mg/kg/h (blinded), in case of shivering episode bolus sodium-chloride (blinded)
  Other Names: Esmeron
  Arms: Rocuronium
Other: placebo — continuous infusion of sodium-chloride (blinded), in case of shivering episode application of rocuronium 0,25mg/kg (blinded)
  Other Names: sodium-chloride
  Arms: Placebo

SUMMARY:
Mild hypothermia improves neurological outcome after cardiac arrest. Neuromuscular blockers are in use, together with analgesia and sedation, during the cooling process in many centers to prevent shivering. Since neuromuscular blockers are accused to be associated with various side effects causing serious harm and/or leading to prolong ICU stay. So economical use seems to be reasonable. Furthermore, the use of neuromuscular blockers may mask epileptic activity. Therefore, post hypoxic seizures might remain undetected.

Aim of this study is to investigate if a continuous application of neuromuscular blockers is necessary to prevent shivering and thereby avoid the counter regulation to achieve the target temperature as soon as possible in mild hypothermic therapy after cardiac arrest.

A single center (university hospital) study. Randomized, double blinded, double dummy study design. Eligible are all adult patients after successful resuscitation due to cardiac arrest of presumed cardiac origin.

All patients receiving mild therapeutic hypothermia after cardiac arrest of presumed cardiopulmonary origin will be included.

Patients <18 years, cardiac arrest >6 hours before admittance at the hospital, patients with known or clinically apparent pregnancy, patients who reach our hospital with a body temperature below 35°C, patients with known allergic reactions against rocuronium, patients with a history of myasthenia gravis, patients with obvious intoxication, wards of the state/prisoners and patients with known epileptic disease will be excluded.

Primary outcome:

Shivering episodes will be scored with the Shivering Assessment Scale.

Secondary outcome:

Total doses of rocuronium, time to target core temperature of 33°C, dissipated energy and total energy needed during the cooling period will be compared between the two groups.

Changes in basal metabolism and depth of relaxation will be ascertained. Furthermore, serum levels of midazolam, fentanyl, rocuronium and stress hormones will be measured.

Train-of-four will be performed to assess the depth of relaxation. Sedation will be monitored via bispectral index; measurement of metabolic activity will be evaluated using indirect calorimetry. Additionally, EEG will be performed to detect epileptiform activities. Blood will be drawn to measure levels of midazolam, fentanyl and rocuronium.

ELIGIBILITY:
Inclusion Criteria:

* all patients receiving mild therapeutic hypothermia after cardiac arrest
* cardiac arrest due to cardiopulmonary origin

Exclusion Criteria:

* patients younger than 18 years
* traumatic cardiac arrest
* cardiac arrest due to exsanguination, strangulation, smoke inhalation, drug overdose, electrocution, hanging or drowning
* known or clinically apparent pregnancy
* no treatment with mild therapeutic hypothermia because of an AND order
* terminal illness
* a body core temperature below 35°C at hospital admission
* known allergic reaction against rocuronium
* history of myasthenia gravis
* obvious intoxication
* ward of the state or prisoner
* known epileptic disease
* cardiac arrest >6 hours prior to hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of shivering episodes | during cooling period (mild therapeutic hypothermia will be performed for 24 hours after cooling initiation, rewarming with 0,4°C per hour until a body core temperature of 36°C is reached); total time of approximately 31 hours
  Shivering episodes will be detected according to the Shivering Assessment Scale

SECONDARY OUTCOMES:
Elapsed time to target temperature | Time from starting the cooling procedure until target temperature is reached - approximately 4 hours after cooling initiation
Dissipated energy to reach the target temperature | Time from starting the cooling procedure until target temperature is reached - approximately 4 hours after cooling initiation
Changes in basal metabolism due to shivering or elevated stress levels | during the first 72 hours after cardiac arrest
Depth of relaxation | during cooling and rewarming period, which will be approximately 30 hours up to 48 hours after initiation of cooling
  via train of four measurement
Changes in serum levels of midazolam, fentanyl and rocuronium | within the first 48 hours of treatment
Number of necessary boli of rocuronium | during colling period (mild therapeutic hypothermia will be performed for 24 hours after cooling initiation, rewarming with 0,4°C per hour until a body core temperature of 36°C is reached); total time of approximately 31 hours
  In case of a shivering episode, a bolus of rocuronium will be administered (0,25mg/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Heidrun Losert, MD, Principal Investigator — Medical University Vienna, Department of Emergency Medicine
Locations (1):
- Medical University of Vienna, Department of Emergency Medicine, Vienna, Vienna, Austria